CLINICAL TRIAL: NCT06746298
Title: A Prospective Study of Expression Profiling-based Assessment of the Efficacy of Neoadjuvant Therapy for Rectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Other Study IDs: RNA-seq-Neo
Record Dates: First submitted 2024-12-17; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Rectal Cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- Rectal cancer patients receiving neoadjuvant therapy

SUMMARY:
This is a prospective study of expression profiling-based assessment of the efficacy of neoadjuvant therapy for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or infertile female
* Patients with rectal adenocarcinoma diagnosed by colonoscopic biopsy
* Neoadjuvant therapy according to guideline recommendations
* Endoscopic biopsy with access to biopsy tissue for subsequent RNA-seq testing
* Patients who do not have a combination of primary malignant tumors elsewhere.
* Patients who understand the purpose of the trial, participate voluntarily and sign an informed consent form.

Exclusion Criteria:

* Samples are not collected, stored, or processed in accordance with specified requirements
* Sample does not meet the requirements for subsequent RNA-seq testing
* Cases enrolled with a subsequent diagnosis other than rectal adenocarcinoma.
* The patient refuses or is unable to complete the entire neoadjuvant treatment
* Lack of post-neoadjuvant imaging results and lack of routine postoperative pathology results.
* Other patients who, in the judgment of the investigator, do not meet the enrollment requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients intended for neoadjuvant therapy
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From the start of the neoadjuvant therapy until just before surgery
  The proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST)

SECONDARY OUTCOMES:
Overall survival | 3 years
  The time from the start of treatment to death due to any cause.
Progression free survival | 3 years
  The period from the date of beginning treatment until the date of disease progression or death from any cause
Total resection rate | One month after surgery
  Surgically removed tissue without residual cancer cells

IPD SHARING:
Plan to Share IPD: Undecided